CLINICAL TRIAL: NCT05637437
Title: Peer-Supported Diabetes Self-Care Intervention to Improve Health Related Quality of Life (HRQoL) and Diabetes Management in Elderly With Type 2 Diabetes (T2DM): A Randomized Control Trial
Brief Title: Peer-Supported Diabetes Self-Care Intervention to Improve Health Related Quality of Life (HRQoL) and Diabetes Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Segufta Dilshad, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GS60104
Record Dates: First submitted 2022-11-12; First posted 2022-12-05 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Elderly; T2DM; HRQoL; Peer Support; Diabetes Management
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants in the control group will receive the usual care of the hospital.
  Interventions: Other: Usual care
- Intervention Group (Experimental): Participants in the intervention group will receive a peer supported diabetes self-care intervention through digital media
  Interventions: Behavioral: Peer supported diabetes self-care intervention; Other: Usual care

INTERVENTIONS:
Behavioral: Peer supported diabetes self-care intervention — Participants in the intervention group will attend a multi-faceted 8 weeks peer supported diabetes self-care intervention through digital communication.
  * Weekly group video telephony meeting facilitated by trained peer supporters.
  * Support and assistance through instant messaging services between peer supporters and participants.
  Arms: Intervention Group
Other: Usual care — Participants in the control group will receive the usual care of the hospital.

SUMMARY:
Diabetes mellitus is the ninth leading cause of mortality worldwide. Diabetes is a chronic condition with a major impact on the life and well-being of individuals, families, and societies globally. The three main types of diabetes are type 1 diabetes mellitus (T1DM), type 2 diabetes mellitus (T2DM), and gestational diabetes mellitus (GDM); approximately 90% of the total cases accounts for T2DM. T2DM is characterized by chronic hyperglycaemia and affects 9.5% of adults aged 20-99 years. The highly burdensome condition is predominantly prevalent in elderly population and distresses 19.3% of elderly aged 65-99 years. Elderly with diabetes have poor Health related Quality of Life (HRQoL) in comparison with their peers of similar age from the general populations.

The determinants of poor HRQoL in elderly with T2DM diabetes population are - poor glycemic control, long duration of diabetes, multiple co-morbidities, depression, high body mass index (BMI), poor self-management practices, higher diabetes related distress, low social support and increased social isolation. Diabetes Self-management Education and Support (DSME/S) is a critical element of care to improve the overall condition of diabetic patients. Self-care does play a critical role in elderly diabetes management. The goal of the current clinical trial is to develop and assess the effectiveness of peer supported diabetes self-care intervention in improving the HRQoL in elderly with type 2 diabetes.

DETAILED DESCRIPTION:
Currently, the prevalence of elderly T2DM in Malaysia is 27.7% compared to 22.7% of 2010. Clinical outcome of diabetes management found deteriorating glycemic control, the mean HbA1c for 2013-2019 ranged from 7.9% - 8.1% and 30.7% of patients achieved the Ministry of Health Diabetes Quality Assurance (QA) target of HbA1c ≤6.5% in 2020. The higher blood sugar level results diabetes complications (cataract 27.2%, neuropathy 45.9% and angina pectoris 18.4%) and poor health related quality of life. Interventions incorporating the cultural, psychosocial, and behavioural factors could improve biophysical, clinical and self-care related outcomes for the elderly with T2DM. People with diabetes require additional resources and support to facilitate and achieve better diabetes HRQoL; and although social and emotional support can occur through family and friends, most people require additional supports from peers.

Peer support refers to the provision of emotional, appraisal and informational support from people who have experiential knowledge of a condition and this support functions to complement, supplement and extend formal primary care services. There is lack of evidence observed on peer supported self-care intervention using 'digital media for the elderly population with T2DM' including appropriate theoretical framework, adequate methodological/designing guidelines and non-pharmacological intervention guideline to improve HRQoL and psychosocial, biomedical and anthropometric outcomes in a single intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age must be 60 years or more
* Diagnosed with T2DM by physician minimum for more than 1 year
* The ability to communicate in Malay or English language properly
* The ability to perform daily activities independently
* No major complications (e.g.- dementia, blind, deaf)
* Planned to continue receiving care at this clinic for next 6 months
* Participated at the usual education session
* Access to a smart phone with internet

Exclusion Criteria:

* Debilitating medical or related condition (e.g. end-stage cancer, severe mental illness)
* Physical inability to provide self-care

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Health Related Quality of Life | Baseline, 3rd and 6th month after intervention
  The HRQoL will be measured by the Revised Version of Diabetes Quality of Life Questionnaire (Bujang et al., 2018). The scale has demonstrated good reliability, composite reliability for each domain was computed as well; "satisfaction" domain showed highest composite reliability of 0.922, followed by "worry" domain (0.794) and "impact" domain (0.781). The range of score for each item is 1 to 5 and total score for the scale is 13 - 65, where higher score indicates poorer quality of life.

SECONDARY OUTCOMES:
Diabetes Self-Care Behavior | Baseline, 3rd and 6th month after intervention
  The Summary of Diabetes Self-Care Activities Scale (Toobert & Glasgow, 1994; Bujang et al., 2016), a 11-item questionnaire measures the frequency of completing different self-care regimen activities over the preceding seven days. All items validated and reliability tested except for smoking status which is in dichotomous response (no/yes). For scoring, general diet = mean number of days for items 1 and 2; specific diet = mean number of days for items 3, and 4, reversing item 4 (0=7, 1=6, 2=5, 3=4, 4=3, 5=2, 6=1, 7=0). Given the low inter-item correlations for this scale, using the individual items is recommended. Exercise = Mean number of days for items 5 and 6; Blood-Glucose Testing = Mean number of days for items 7 and 8; Foot-Care = Mean number of days for items 9 and 10; Smoking Status = Item 11 (0 = non-smoker, 1 = smoker), and number of cigarettes smoked per day.
Social Support | Baseline, 3rd and 6th month after intervention
  Social Support will be measured using the Malay version of Medical Outcomes Study Social Support Survey, which consists of four dimensions/subscales (emotional, tangible support, positive social interaction and affectionate support) and 19 items (Norhayati et al., 2015). Both the English and the Malay versions has good reliability (α= 0.91 and α=0.96 respectively). Responses were summed to create a total score ranging from 0 to 100, with the higher score indicating greater outcome expectations. Scores were rescaled to a 0 to 100 on a ratio scale, with higher scores indicating a higher social support. The original instrument showed acceptable reliability (α > 0.91).
Self-Efficacy | Baseline, 3rd and 6th month after intervention
  Self-efficacy will be measured by the the Diabetes Empowerment Scale, which is a 8-item short form of questionnaire, measures the psychosocial self-efficacy of people with diabetes (Anderson et al., 2003) and evaluate the empowerment levels of individuals in relation to their state of health. The result of the scale obtains by the average of the sum of all included items, in which higher values are related to higher perceptions of psychosocial self-efficacy. The coefficient of Cronbach's alpha of 0.84 was obtained and the unidimensional nature of the scale was confirmed.
Depression | Baseline, 3rd and 6th month after intervention
  The Malay Version Brief Patient Health Questionnaire (Shaaban, 2005) is a 9-item depression scale measures the level of depression. Each question has scale from 0-3 reflecting the severity of the symptoms. The possible total score ranges from 0-27. The total score greater than 10 had a sensitivity and specificity of 88% for major depressive disorder. Reliability and validity of the scale has indicated a sound psychometric property with high internal consistency. Scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively.
HbA1c level | Baseline, 3rd and 6th month after intervention
  Electronic medical record of the hospital
Lipid Profiles | Baseline, 3rd and 6th month after intervention
  Electronic medical record of the hospital
Body Mass Index | Baseline, 3rd and 6th month after intervention
  Electronic medical record of the hospital
Systolic and Diastolic Blood Pressure | Baseline, 3rd and 6th month after intervention
  Electronic medical record of the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr Sazlina S Ghazali, MBBS, PhD, Study Chair — University Putra Malaysia; A/Prof. Cheong Ai Theng, MBBS, PhD, Study Director — University Putra Malaysia; Segufta Dilshad, EMPH, Principal Investigator — University Putra Malaysia
Locations (1):
- Universiti Putra Malaysia (UPM), Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AADE. AADE7 Self-Care Behaviors. Diabetes Educ. 2008 May-Jun;34(3):445-9. doi: 10.1177/0145721708316625. No abstract available. PMID 18535317
- [Background] Andreae SJ, Andreae LJ, Richman JS, Cherrington AL, Safford MM. Peer-Delivered Cognitive Behavioral Training to Improve Functioning in Patients With Diabetes: A Cluster-Randomized Trial. Ann Fam Med. 2020 Jan;18(1):15-23. doi: 10.1370/afm.2469. PMID 31937528
- [Background] Castillo-Hernandez KG, Laviada-Molina H, Hernandez-Escalante VM, Molina-Segui F, Mena-Macossay L, Caballero AE. Peer Support Added to Diabetes Education Improves Metabolic Control and Quality of Life in Mayan Adults Living With Type 2 Diabetes: A Randomized Controlled Trial. Can J Diabetes. 2021 Apr;45(3):206-213. doi: 10.1016/j.jcjd.2020.08.107. Epub 2020 Sep 2. PMID 33129754
- [Background] Ghasemi M, Hosseini H, Sabouhi F. Effect of Peer Group Education on the Quality of Life of Elderly Individuals with Diabetes: A Randomized Clinical Trial. Iran J Nurs Midwifery Res. 2019 Jan-Feb;24(1):44-49. doi: 10.4103/ijnmr.IJNMR_39_17. PMID 30622577
- [Background] Oluchi SE, Manaf RA, Ismail S, Kadir Shahar H, Mahmud A, Udeani TK. Health Related Quality of Life Measurements for Diabetes: A Systematic Review. Int J Environ Res Public Health. 2021 Sep 1;18(17):9245. doi: 10.3390/ijerph18179245. PMID 34501838
- [Background] Peimani M, Monjazebi F, Ghodssi-Ghassemabadi R, Nasli-Esfahani E. A peer support intervention in improving glycemic control in patients with type 2 diabetes. Patient Educ Couns. 2018 Mar;101(3):460-466. doi: 10.1016/j.pec.2017.10.007. Epub 2017 Oct 12. PMID 29055655
- [Background] Sazlina SG, Zaiton A, Nor Afiah MZ, Hayati KS. Predictors of health related quality of life in older people with non-communicable diseases attending three primary care clinics in Malaysia. J Nutr Health Aging. 2012 May;16(5):498-502. doi: 10.1007/s12603-012-0038-8. PMID 22555798
- [Background] Seah SJ, Zheng H, Lim RBT. Efficacy of community-based self-care interventions to improve biophysical, psychosocial or behavioural outcomes among community-dwelling older adults with type 2 diabetes: A systematic review and meta-analysis. Diabetes Res Clin Pract. 2020 Nov;169:108411. doi: 10.1016/j.diabres.2020.108411. Epub 2020 Sep 6. PMID 32898575
- [Background] Shahsavari A, Estebsari F, Atashzadeh-Shoorideh F, Ilkhani M. The effect of peer support on quality of life among type 2 diabetic patients in deprived areas in Iran: A randomized clinical trial. J Educ Health Promot. 2021 Sep 30;10:345. doi: 10.4103/jehp.jehp_72_21. eCollection 2021. PMID 34761031
- [Background] Ahmad Sharoni SK, Abdul Rahman H, Minhat HS, Shariff-Ghazali S, Azman Ong MH. The effects of self-efficacy enhancing program on foot self-care behaviour of older adults with diabetes: A randomised controlled trial in elderly care facility, Peninsular Malaysia. PLoS One. 2018 Mar 13;13(3):e0192417. doi: 10.1371/journal.pone.0192417. eCollection 2018. PMID 29534070
- [Background] Teare MD, Dimairo M, Shephard N, Hayman A, Whitehead A, Walters SJ. Sample size requirements to estimate key design parameters from external pilot randomised controlled trials: a simulation study. Trials. 2014 Jul 3;15:264. doi: 10.1186/1745-6215-15-264. PMID 24993581
- [Background] Sinclair A, Saeedi P, Kaundal A, Karuranga S, Malanda B, Williams R. Diabetes and global ageing among 65-99-year-old adults: Findings from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2020 Apr;162:108078. doi: 10.1016/j.diabres.2020.108078. Epub 2020 Feb 14. PMID 32068097
- See also: Institute for Public Health 2020. National Health and Morbidity Survey (NHMS) 2019: Non-communicable diseases, healthcare demand, and health literacy-Key Findings — https://iptk.moh.gov.my/images/technical_report/2020/4_Infographic_Booklet_NHMS_2019_-_English.pdf
- See also: World Health Organization. (2015). World report on ageing and health. World Health Organization. — https://apps.who.int/iris/handle/10665/186463